CLINICAL TRIAL: NCT05126862
Title: Measurement and Modification of Threat Interpretation Bias in Neurodegenerative Movement Disorders (Aims 2 & 3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jessie Gibson, PhD, RN, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR 210113; KL2TR003016 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease; Parkinson Disease
Keywords: Anxiety; Interpretation bias; Cognitive bias modification
MeSH Terms: conditions — Huntington Disease; Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two single groups will be recruited: one including participants with Huntington's disease and the other including participants with Parkinson's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MindTrails pilot (Experimental): This intervention involves completion of five, 20-minute MindTrails online training sessions over five weeks.
  Interventions: Behavioral: MindTrails

INTERVENTIONS:
Behavioral: MindTrails — MindTrails is a web-based cognitive bias modification intervention. Training sessions are designed to encourage cognitive flexibility through repeated practice assigning benign resolutions to ambiguous, anxiety-provoking situations.

SUMMARY:
The purpose of this study is conduct a pilot open trial of a web-based cognitive bias modification intervention to reduce anxiety symptoms in persons with Huntington's disease and persons with Parkinson's disease.

DETAILED DESCRIPTION:
After being informed about the study and giving informed consent, participants will enroll in a pilot open trial of MindTrails, a web-based cognitive bias modification intervention. Participants will complete five, 20-minute MindTrails training sessions over five weeks. Additionally, assessments of anxiety, interpretation bias, and other related outcomes will be completed at baseline, week 3, week 5, and 2 months following the last training session. Participants will each complete a semi-structured interview to provide qualitative feedback about their experiences with MindTrails and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Huntington's disease or Parkinson's disease
* Age 21 or older
* Has anxiety symptoms (NeuroQoL Anxiety short form >12)

Exclusion Criteria:

* Unable to read and understand English
* Previously diagnosed with dementia
* Not located in the USA

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie S Gibson, PhD, RN, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: MindTrails Pilot in Parkinson's Disease; Experimental: MindTrails Pilot in Huntington's Disease: This intervention involves completion of five, 20-minute MindTrails online training sessions over five weeks.
Period: Overall Study
Arm/Group | Experimental: MindTrails Pilot in Parkinson's Disease | Experimental: MindTrails Pilot in Huntington's Disease
Started | 22 | 21
Completed | 14 | 12
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: MindTrails Pilot in Parkinson's Disease | Experimental: MindTrails Pilot in Huntington's Disease | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.05 (11.20) | 48.95 (11.81) | 56.67 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 13 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43
Education [Count of Participants; unit: Participants]
  High School | 2 | 3 | 5
  Some College | 3 | 9 | 12
  Associate's Degree | 4 | 1 | 5
  Bachelor's | 6 | 6 | 12
  Master's | 4 | 1 | 5
  Doctorate/PhD | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Completing at Least 50% of the MindTrails Sessions
Description: Proportion of participants completing at least 50% of the MindTrails sessions (defined as proportion of participants who completed outcome assessments for at least 2 of the 3 timepoints measured during the intervention: baseline, week 3, and week 5)
Time Frame: Between baseline and week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: MindTrails Pilot in Parkinson's Disease | Experimental: MindTrails Pilot in Huntington's Disease
Number analyzed (Participants) | 22 | 21
Participants | 14 | 14

2. Primary Outcome: Participant Perceptions of Perceived Benefits and Limitations of MindTrails
Description: All participants in each arm were invited to complete a semi-structured interview to assess their experience with the intervention or barriers to beginning or completing the intervention. Interviews were transcribed, and separate codebooks were developed for PD and HD transcripts. Each transcript was coded by 2 coders, and any disagreements were resolved by a third coder. Frequency of overlapping codes under the "Experiences completing MindTrails" theme for each group (PD and HD) are reported here.
Time Frame: After completion of the intervention (week 5)
Population: All participants in each arm were invited to complete a semi-structured interview; 14 PD participants and 10 HD participants completed interviews.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: MindTrails Pilot in Parkinson's Disease; Experimental: MindTrails Pilot in Huntington's Disease: This intervention involves completion of five, 20-minute MindTrails online training sessions over five weeks. Participants were invited to complete an interview about their experience with the intervention and/or barriers to completion.
Arm/Group | Experimental: MindTrails Pilot in Parkinson's Disease | Experimental: MindTrails Pilot in Huntington's Disease
Number analyzed (Participants) | 14 | 10
Participants
  did not need help to complete | 12 | 9
  needed caregiver assistance | 1 | 1
  completed it on phone | 3 | 1
  completed on computer | 3 | 3
  participant baseline characteristics influence experience positively | 4 | 4
  participant baseline characteristics influence experience negatively | 4 | 5
  positive experience/ enjoyed MindTrails | 7 | 4
  easy to navigate/ straight-forward | 13 | 10
  interesting/ engaging | 5 | 2
  neutral experience with MindTrails | 2 | 2
  did not enjoy MindTrails | 0 | 1
  difficulty with and/or did not like forced response choice | 5 | 3
  redundancy | 4 | 2

ADVERSE EVENTS:
Time Frame: Approximately 13 weeks (5 week intervention period and 2 month follow-up).
Description: Because this study posed minimal risk to the subject, adverse events were only to be collected or recorded if a causal relationship to the study intervention was suspected. No adverse events were reported during the course of the study.
Arm/Group | Experimental: MindTrails Pilot in Parkinson's Disease | Experimental: MindTrails Pilot in Huntington's Disease
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT05126862/Prot_SAP_000.pdf